CLINICAL TRIAL: NCT06684756
Title: The Comparison of the Efficacy and Safety of Vacuum-Assisted and Conventional Ureteral Access Sheath in Retrograde Intrarenal Surgery: A Randomized Controlled Prospective Multicenter Study
Brief Title: Comparison of Vacuum-Assisted and Conventional Ureteral Access Sheath in Retrograde Intrarenal Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Mehmet Fatih Şahin, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024.288.10.16
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Kidney Calculi; Kidney Stones
Keywords: kidney stone; retrograde intrarenal surgery; ureteral access sheath; vacuum assisted
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with conventional UAS being used in their RIRS operations (Active Comparator): The patient population will be selected from cases determined by randomization and used with UAS without an aspiration (conventional) during RIRS.
  Interventions: Procedure: Retrograde intrarenal surgery
- Patients with vacuum assisted UAS being used in their RIRS operations (Experimental): The patient population will be selected from cases determined by randomization and used with UAS with an aspiration and flexible tip, different from the conventional one during RIRS.
  Interventions: Procedure: Retrograde intrarenal surgery

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery — Flexible optic devices and lasers fragment kidney stones during this operation. In this surgery, an ureteral access sheath is recommended to be used.

SUMMARY:
This study aims to compare the efficacy and safety, the ratio of stone-free rates, and complications of two types of access sheaths used in retrograde intrarenal surgery to treat upper urothelial stones. The access sheath types are those with vacuum aspiration and the conventional ones.

DETAILED DESCRIPTION:
The use of ureteral access sheath (UAS) during Retrograde Intrarenal Surgery (RIRS) has been proven effective and reliable in recent years, and publications indicate that it reduces stone-free rates (SFR). Their use is also recommended in the European Urology Guidelines because it improves image quality, reduces intrarenal pressure, and shortens the operation time. For this reason, it has been routinely used in many RIRS cases. In cases where non-vacuum-assisted UAS is used, fragments during stone fragmentation remain in the kidney, and since it is not possible to remove the stones simultaneously, the image may be distorted, and the operation duration may be prolonged. All these may pave the way for postoperative infectious complications. In addition to non-vacuum-assisted UAS, new UASs with flexible ends and vacuum-assisted aspiration have been introduced in the last few years (ClearPetra). Thanks to the aspiration connected to the system, stone fragments can be removed from the body with negative pressure during stone fragmentation. Continuous circulation prevents bleeding during fragmentation and blurring of the visual field due to stone fragments. In addition, since the stone fragments pass through the edges of the sheath without breaking and are removed, a perfect field of view can be provided. Unlike the classical UAS, the tip is flexible, allowing for the safe removal of lower pole stones. Many studies in the literature compare the success and complications of RIRS in cases where conventional UAS was used and not used. In addition, there are publications related to using the newly introduced aspiration access sheath in percutaneous nephrolithotomy. In retrospective publications on using this UAS in RIRS, it has been shown that stone-free rates, operation time, hemoglobin loss, and postoperative infective complications are more successful on the 1st and 30th postoperative days compared to cases where non-vacuum-assisted UAS was used. There is no randomized controlled prospective publication on this subject. This study aims to compare the complications and stone-free rates of RIRS cases where non-vacuum-assisted UAS and new vacuum-assisted UAS were used.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients below 85 years of age
* Patients with 11-13 FR conventional/vacuum-assisted ureteral access sheath (UAS) during retrograde intrarenal surgery

Exclusion Criteria:

* Patients with non-sterile preoperative urine culture
* Patients with renal anatomic anomalies
* Patients with a solitary (single) kidney
* Patients with insufficient data
* Patients under the age of 18, above the age of 85
* Patients without an UAS during RIRS
* Patients without 11-13Fr UAS during RIRS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rates | Stone-free status will be checked by performing a non-contrast abdominal CT scan 1 month after the operation.
  Presence/absence of residual fragments in postoperative imaging, if any, diameter of longest axis in mm.

SECONDARY OUTCOMES:
Complication rates | Peroperative complication rates will be determined during the operation, and postoperative complications will be re-evaluated during hospitalization before discharge or in the first month after discharge.
  Peroperative and postoperative complication rates, whether UAS related or not

CONTACTS AND LOCATIONS:
Overall Officials: Cenk M. Yazici, Professor, Study Director — Namik Kemal University
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Xu Y, Liu Z, Liang J, Lai D, Guan W, Xu G. Using vacuum-assisted ureteral access sheath in the treatment of complex steinstrasse. Urolithiasis. 2023 Jun 22;51(1):89. doi: 10.1007/s00240-023-01462-2. PMID 37347309
- [Background] Zhang Z, Xie T, Li F, Wang X, Liu F, Jiang B, Zou X, Zhang G, Yuan Y, Xiao R, Wu G, Qian B. Comparison of traditional and novel tip-flexible suctioning ureteral access sheath combined with flexible ureteroscope to treat unilateral renal calculi. World J Urol. 2023 Dec;41(12):3619-3627. doi: 10.1007/s00345-023-04648-w. Epub 2023 Oct 11. PMID 37821778
- [Background] Nao T, Iga R, Yoshimura R, Kurano Y, Yamamoto S, Tamura K. A new method for effective use of the ClearPetra ureteral access sheath for a giant ureteral stone. Urol Case Rep. 2023 Oct 23;51:102599. doi: 10.1016/j.eucr.2023.102599. eCollection 2023 Nov. PMID 38024505
- [Result] Gauhar V, Traxer O, Castellani D, Sietz C, Chew BH, Fong KY, Hamri SB, Gokce MI, Gadzhiev N, Galosi AB, Yuen SKK, El Hajj A, Ko R, Zawadzki M, Sridharan V, Lakmichi MA, Corrales M, Malkhasyan V, Ragoori D, Soebhali B, Tan K, Chai CA, Tursunkulov AN, Tanidir Y, Persaud S, Elshazly M, Kamal W, Tefik T, Shrestha A, Tiong HC, Somani BK. Could Use of a Flexible and Navigable Suction Ureteral Access Sheath Be a Potential Game-changer in Retrograde Intrarenal Surgery? Outcomes at 30 Days from a Large, Prospective, Multicenter, Real-world Study by the European Association of Urology Urolithiasis Section. Eur Urol Focus. 2024 Dec;10(6):975-982. doi: 10.1016/j.euf.2024.05.010. Epub 2024 May 24. PMID 38789313